CLINICAL TRIAL: NCT03153540
Title: A Randomized, Double-blinded, Sham-controlled Cross-over Study of Theta-burst Transcranial Magnetic Stimulation in Nonfluent/Agrammatic Variant Primary Progressive Aphasia
Brief Title: Transcranial Magnetic Stimulation in Nonfluent/Agrammatic Variant Primary Progressive Aphasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H16-01327
Record Dates: First submitted 2017-03-01; First posted 2017-05-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Primary Progressive Nonfluent Aphasia
Keywords: Aphasia; Agrammatism; Frontotemporal Dementia; Tauopathies; Neurodegenerative Diseases; Language Disorders; Frontotemporal Lobar Degeneration
MeSH Terms: conditions — Primary Progressive Nonfluent Aphasia; Aphasia; Aphasia, Broca; Frontotemporal Dementia; Tauopathies; Neurodegenerative Diseases; Language Disorders; Frontotemporal Lobar Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active iTBS (Active Comparator): Device: MagPro X100 stimulator equipped with the B65 fluid-cooled coil for dominant Inferior Frontal Gyrus (IFG) stimulation (MagPro, Medtronic).
  Intervention: 10 sessions daily of iTBS over 2 weeks. Active-iTBS consists of intermittent Theta Burst Stimulation to the dominant IFG (120% of resting motor threshold, bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz for 600 pulses total over 3 min).
  Interventions: Device: Active iTBS
- Sham iTBS (Sham Comparator): Device: MagPro X100 stimulator applied to dominant inferior frontal lobe.
  Intervention: 10 sessions daily of sham iTBS over 2 weeks. Sham sessions involve a click replicating the sound of the magnetic discharge, without any magnetic pulse being delivered.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Active iTBS — Intermittent theta burst transcranial magnetic stimulation
  Arms: Active iTBS
Device: Sham iTBS — Sham intervention
  Arms: Sham iTBS

SUMMARY:
Nonfluent/agrammatic variant primary progressive aphasia (nf/avPPA) is a fatal neurodegenerative disease that begins with isolated language deficits. There is currently no cure or treatment for this disease. Repetitive Transcranial Magnetic Stimulation (rTMS), a noninvasive neuromodulatory technique, is effective in major depression, and studied in many other conditions including nf/avPPA. Here the investigators propose to study the feasibility and change in language and brain function of a newer rTMS protocol (intermittent theta-burst stimulation, iTBS) using a randomized, blinded crossover design: participants will receive active or sham iTBS for two weeks and then switch groups without them or clinicians knowing their group. The investigators hypothesize that brain function and performance with language tasks will change after active iTBS.

DETAILED DESCRIPTION:
This study is a randomized controlled blinded cross-over treatment trial that involves 20 iTBS treatment sessions (10 active treatment sessions; 10 sham treatment sessions) and the study will last between 6 weeks. There will be 20 treatment visits (Monday-Friday) each lasting 10-40 minutes. Whether the participant is randomly assigned to active or sham treatment, the participant will receive daily 10 minute session of iTBS treatment. Some sessions will include behavioral and neurophysiological measures.

In addition, participants will complete cognitive testing, and neuro-imaging, including functional magnetic resonance (fMRI), functional near infrared spectroscopy (fNIRS) and electroencephalography (EEG) prior to the commencement of iTBS/sham treatment and at post-treatment. Safety and tolerability will be evaluated during daily iTBS treatments.

After 10 iTBS treatment visits over 2 weeks, a clinical assessment will be done to see if the participants are responding to the iTBS treatment with a targeted language assessment and neuro-imaging as described above. After 2 weeks of "wash-out", where the subjects do not receive any treatments, the participants will undergo another 2 weeks of iTBS treatment. On the first iTBS session after the 2-week washout period, participants will undergo a targeted language assessment and EEG/fNIRS. At the final iTBS session at 6 weeks, subjects will again undergo a targeted language assessment, EEG/fNIRS, and fMRI. At that point, after 6 weeks, the cross-over study is finished.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with nonfluent-agrammatic variant primary progressive aphasia (nfvPPA), by 2011 Gorno-Tempini diagnostic criteria.
* Frontotemporal lobar degeneration modified clinical dementia rating scale (FTLD-CDR) score ≤4 (mild).
* Is voluntary and competent to consent to treatment, or if demented, to assent and co-consent can be obtained by their legal next-of-kin, legal guardian, or substitute decision maker.
* Speaks English enough to be able to complete neuropsychological testing.
* Able to adhere to the treatment schedule.
* Has a study partner available to answer the Progressive Aphasia Severity Scale (PASS) questionnaire.

Exclusion Criteria:

* Uncorrected visual or hearing impairment by self report.
* History of substance dependence or abuse within the last 3 months.
* Has active suicidal intent.
* Has a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of major depressive disorder, bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
* Concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump.
* Any significant neurological disorder other than nfvPPA including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, history of epilepsy, known cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes in the previous 6 months.
* Is currently (or in the last 4 weeks) taking lorazepam greater than 2 mg daily (or equivalent) or any dose of an anticonvulsant, due to the potential to limit rTMS efficacy.

Exclusion Criteria for TMS Participation:

- Does not pass the TMS adult safety screening (TASS) questionnaire (e.g. has an intracranial implant)

Exclusion Criteria for MRI Participation:

* Severe claustrophobia.
* Cardiac pacemakers or ferromagnetic implants.
* Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 6 weeks
  Safety will be measured by incidence of treatment-emergent adverse events
Tolerability levels according to the daily Comfort Rating Questionnaire (CRQ) | 6 weeks
  Tolerability will be measured by daily Comfort Rating Questionnaire (CRQ) between sham and active interventions and compared using Chi-square. A mean score across all treatment sessions above 6 on more than 2 items on the CRQ will be considered as severe. A mean score across all treatment sessions between 4 and 6 on more than 2 items on the CRQ will be considered as moderate tolerability. A mean score across all treatment sessions below 4 on the majority of items will be considered as mild tolerability.
Drop out rate | 6 weeks
  Feasibility will be measured by drop out rate. A drop out rate >50% will be considered as an indication of non-feasibility of current protocol.

SECONDARY OUTCOMES:
Changes in the Verb and Object Naming Test score | 6 weeks
  Verb and Object Naming Test score at baseline and at 2, 4, and 6 weeks
Changes in the Make a Sentence Test score | 6 weeks
  Make a Sentence Test score at baseline and at 2, 4, and 6 weeks
Changes in the Sentence Comprehension Test score | 6 weeks
  Sentence Comprehension Test score at baseline and at 2, 4, and 6 weeks
Changes in the Apraxia of Speech Rating Scale score | 6 weeks
  Apraxia of Speech Rating Scale score at baseline and at 6 weeks
Changes in the Clinical Global Impression of Change score | 6 weeks
  Clinical Global Impression of Change score at baseline and at 2, 4, and 6 weeks
Changes in the Progressive Aphasia Severity Scale rating | 6 weeks
  Progressive Aphasia Severity Scale rating at baseline and at 6 weeks
Changes in the Western Aphasia Battery rating | 6 weeks
  Western Aphasia Battery rating at baseline and at 6 weeks
Changes in the Montreal Cognitive Assessment Battery score | 6 weeks
  Montreal Cognitive Assessment Battery score at baseline and at 6 weeks
Changes in the Frontal Assessment Battery score | 6 weeks
  Frontal Assessment Battery score at baseline and at 6 weeks
Changes in the whole-brain functional connectivity measured using functional Magnetic Resonance Imaging (MRI) | 6 weeks
  fMRI at baseline and at 2 and 6 weeks
Changes in the brain cortical blood oxygenation measured using functional Near Infrared Spectroscopy (fNIRS) | 6 weeks
  fNIRS at baseline and at 2, 4, and 6 weeks
Changes in the brain cortical electrical activity measured using quantitative electroencephalography (EEG) | 6 weeks
  EEG at baseline and at 2, 4, and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, Principal Investigator — University of British Columbia
Locations (1):
- Non-Invasive Neurostimulation Therapies lab, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No